CLINICAL TRIAL: NCT01104831
Title: The Efficacy and Cost Effectiveness of Preoperative and Postoperative Cryotherapy in Proximal Tibia Fractures
Acronym: ARCTIC CAT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inadequate recruitment.
Sponsor: University of Manitoba (Other)
Collaborators: Orthopedic Research and Education Foundation (Other); Orthopedic Trauma Association (Unknown)
Responsible Party: Jesse Shantz, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2009:035
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2011-04

CONDITIONS: Proximal Tibia Fracture
Keywords: Tibial Plateau Fracture; AO/OTA 41
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 21 degree Cooling (Placebo Comparator): Room temperature water circulated through cryotherapy sleeve.
  Interventions: Device: Room temperature cuff
- 10 degree cooling (Active Comparator): Cooled water circulated through a cryotherapy sleeve.
  Interventions: Device: Cryotherapy

INTERVENTIONS:
Device: Cryotherapy — cooled sleeve placed over fracture site.
  Arms: 10 degree cooling
Device: Room temperature cuff — sleeve with room temperature water placed over fracture site.
  Arms: 21 degree Cooling

SUMMARY:
Consenting patients with proximal tibia fractures will be randomized to 10 degree or 21 degree cryotherapy sleeves. Time to discharge and complications will be monitored.

Primary outcome measure: Cost of Treatment (based on length of stay) Secondary outcome measures: Satisfaction/pain relief and narcotic requirement

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Trauma patients with single-system musculoskeletal injuries.
* Proximal tibia fractures treated with open reduction and internal fixation.
* Unilateral proximal tibial injuries.

Exclusion Criteria:

* Previous ipsilateral knee surgery
* Upper extremity injuries impairing mobilization
* Pre-existing ipsilateral neurologic condition or acute ipsilateral neurologic injury
* Associated injuries impairing mobilization
* Suspected or confirmed compartment syndrome
* Open fractures
* Patients previously on narcotics
* Patients with impaired sensorium Concurrent head injury Intoxication

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cost | 3 months

SECONDARY OUTCOMES:
VAS Pain Score | 2 weeks
Narcotic Requirements | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jesse A Shantz, MD, MBA, Principal Investigator — University of Manitoba
Locations (1):
- Winnipeg Health Sciences Centre, Winnipeg, Manitoba, Canada